CLINICAL TRIAL: NCT00861042
Title: An Open-label follow-on Trial to Assess the Long-term Safety and Efficacy of Oral SPM 927 in Subjects With Diabetic Neuropathy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: UCB Pharma (Industry)
Responsible Party: Study Director, UCB
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SP0665
Record Dates: First submitted 2009-03-12; First posted 2009-03-13 (Estimated); Last update posted 2024-01-29 (Actual); Status verified 2024-01

CONDITIONS: Painful Diabetic Neuropathy
Keywords: Lacosamide, Vimpat®
MeSH Terms: conditions — Diabetic Neuropathies | interventions — 2-(acetylamino)-3-methoxy-N-(phenylmethyl)-, (2R)-; Lacosamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental)
  Interventions: Drug: SPM927/Lacosamide

INTERVENTIONS:
Drug: SPM927/Lacosamide — SPM927 (film-coated tablets, 25/50/100mg per tablet), dosage up to 400mg/day, intake in the morning and in the evening; duration of intake depending on individual trial participation SPM927 (film-coated tablets, 25/50/100mg per tablet), dosage up to 400mg/day, intake in the morning and in the evening; duration of intake depending on individual trial participation
  Other Names: SPM927 / Lacosamide / Vimpat®

SUMMARY:
The primary objective of the trial is to assess the tolerability and safety of long-term SPM 927 administration in subjects with diabetic neuropathy.

ELIGIBILITY:
Inclusion Criteria:

* Subject has successfully completed a previous trial with SPM 927 in diabetic neuropathy and, in the investigator's opinion, would benefit from long-term administration of SPM 927.
* Subject has stable, good or fair diabetic control (HbA1c ≤10% ).

Exclusion Criteria:

* Subject has other conditions that cause neuropathic pain at least as severe as the diabetic pain, i.e. peripheral arterio-vascular disease.
* Subject receives treatment for seizures.
* Subject has had an amputation related to diabetes, other than toe amputation.
* Subject has major skin ulcers.
* Subject has clinically significant ECG abnormalities.
* Subject expects to take during the study: TCAs, mexiletine hydrochloride, lidoderm patch, tramadol, AEDs, dextromethorphan, opioids, capsaicin, skeletal muscle relaxants, benzodiazepines or over-the-counter medications with centrally acting properties.
* Subject has laboratory values which are outside the normal range and judged by the investigator to be clinically significant.
* Subject has liver function tests (AST, ALT, alkaline phosphatase, total bilirubin, or GGT) ≥ 2x ULN at Visit 1.
* At Visit 1, subject has impaired renal function, i.e., creatinine clearance (ClCr) is lower than 60 mL/min.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 69 (Actual)
Dates: Start 2002-04; Primary Completion 2004-12 (Actual); Study Completion 2005-03 (Actual)

PRIMARY OUTCOMES:
Assess the tolerability and safety of long-term SPM 927 administration in subjects with diabetic neuropathy | Assessments during whole course of the trial: spontaneously by the subject and observed by the investigators during site visits
Adverse events reported spontaneously by the subject or observed by the investigator | Assessments during whole course of the trial: spontaneously by the subject and observed by the investigators during site visits.
Changes laboratory, ECG and vital signs parameters. | Assessments during whole course of the trial: spontaneously by the subject and observed by the investigators during site visits.
Changes in physical or neurological examination findings | Assessments during whole course of the trial: spontaneously by the subject and observed by the investigators during site visits.
Subject withdrawal due to adverse events | Assessments during whole course of the trial: spontaneously by the subject and observed by the investigators during site visits.

SECONDARY OUTCOMES:
The secondary objective is to gather further information on the efficacy of SPM 927 in this indication. | Daily assessment during entire trial participation including assessments at site visits
Within-subject change in average pain score: Daily assessments throughout the trial | Daily assessment during entire trial participation including assessments at site visits
Change in subject's perception of different neuropathic pain qualities during specific site visit | Daily assessment during entire trial participation including assessments at site visits
Time to exit (days) de to lack of efficacy of treatment | Daily assessment during entire trial participation including assessments at site visits
Change in subject's perception of sleep and activity throughout the trial, daily assessments | Daily assessment during entire trial participation including assessments at site visits
Patient's Global Impression of Change in Pain (PGIC) during specific site visit | Daily assessment during entire trial participation including assessments at site visits
Clinical Global Impression of Change in Pain (CGIC): Assessments during specific site visit | Daily assessment during entire trial participation including assessments at site visits
Quality of life assessments during specific site visits | Daily assessment during entire trial participation including assessments at site visits

CONTACTS AND LOCATIONS:
Overall Officials: UCB Clinical Trial Call Center, Study Director — +1 877 822 9493 (UCB)

REFERENCES:
- [Result] Shaibani A, Biton V, Rauck R, Koch B, Simpson J. Long-term oral lacosamide in painful diabetic neuropathy: a two-year open-label extension trial. Eur J Pain. 2009 May;13(5):458-63. doi: 10.1016/j.ejpain.2008.05.016. Epub 2008 Jul 10. PMID 18619874